CLINICAL TRIAL: NCT00262158
Title: The Survey of Cigarette Consumption
Brief Title: Analysis of 'Tobacco and Alcohol Tax Law' and Its Impact on Cigarette Consumption
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Bureau of Health Promotion,DoH,Taiwan (Unknown)
Other Study IDs: EC 0930704
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2005-12-06 (Estimated); Status verified 2005-12

CONDITIONS: Smoking Status; Cigarette Consumption
Keywords: smoking status; cigarette consumption

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
This project is the survey on smoking behavior in Taiwan. The survey information will be used to analyze the influence of the earmarked tax of cigarettes on (1)the consumption of cigarette,(2)the substitution between the consumption of domestic and imported cigarettes, and(3)the consumption of other addictive goods.

DETAILED DESCRIPTION:
The specific aims of this study are as follows:

Test hypotheses regarding the influence of cigarette tax on the consumption of cigarette and other addictive goods:

To test the hypothesis that the imposition of earmarked tax of cigarettes will cause decrease of cigarette consumption.

To test the hypothesis that the imposition of earmarked tax of alcohol will cause the substitution of consumption of domestic and imported cigarettes.

To test the hypothesis that the imposition of earmarked tax of cigarettes will cause the substitution of consumption of high-priced and low-priced cigarettes.

To test the hypothesis that the imposition of earmarked tax of cigarettes will cause decrease of the consumption of other addictive goods.

To test the hypothesis that the imposition of earmarked tax of alcohol will cause decrease of alcohol consumption.

To test the hypothesis that the imposition of earmarked tax of alcohol will cause decrease of the consumption of other addictive goods.

To test the hypothesis that price effect of earmarked cigarette tax on addicted smokers is less than on non-addicted smokers.

To test the hypothesis that price effect earmarked cigarette tax on heavy smokers is less than on light and moderate smokers.

To test the hypothesis that earmarked cigarette tax and alcohol tax are regressive.

Test hypotheses regarding the influence of information, knowledge attitude on cigarette smoking and smoking cessation.

To test the hypothesis that exposure to anti-smoking information is negatively related to cigarette smoking and positively related to smoking cessation.

To test the hypothesis that exposure to information on cigarette promotion is positively related to cigarette smoking and negatively related to smoking cessation.

To test the hypothesis that people perceiving high risk of cigarette smoking are less likely to smoke.

To test the hypothesis that highly risk averse people are less likely to smoke.

ELIGIBILITY:
Inclusion Criteria:

- The random sample of population over 18 years old.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4000
Dates: Start 2004-08; Study Completion 2004-09

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Wen Ysai, Ph.D., Principal Investigator — NHRI